CLINICAL TRIAL: NCT00288990
Title: Impact of Neutralizing Antibodies on Interferon Responsive Genes Highlights Biomarker Response.
Brief Title: A Serologic Study to Correlate Beta-IFN NAb Titers to Beta-IFN Induced Biomarker Response in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Other Study IDs: 008-05-AVX
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: subjects who are NAb positive
- 2: Subjects who are antibody negative
- 3: subjects who are BAb positive

SUMMARY:
Study Title: A Serologic Study to Correlate b-IFN NAb titers to b-IFN Induced Biomarker Response in Patients with Multiple Sclerosis

Objectives: Subjects currently on any of the three b-IFN preparations (Avonex (Interferon b-1a 30 mcg IM Q 7 days), Rebif (Interferon b-1a 22 or 44mcg SC TIW), or Betaseron (Interferon b-1b 250mcg SC QOD)) will be enrolled to one of 3 groups:

Group 1: Approximately 200 subjects will be enrolled who are NAb+ (titer ³ 20NU/ml) Group 2: Approximately 50 subjects will be enrolled who are BAb- (titer <8U) and NAb- (titer <20 NU/ml) Group 3: Approximately 50 subjects will be enrolled who are BAb+ (titer ³8U) and NAb- (titer <20 NU/ml)

The primary objective of this study is to compare baseline b-IFN induced MxA mRNA response in neutralizing antibody positive (NAb+, titers ³ 20NU/ml, Group 1) vs. antibody negative (NAb-, titers < 20NU/ml, BAb-, titers <8U, Group 2) patients.

Secondary objectives are:

1. To compare b-IFN induced MxA mRNA response in neutralizing antibody positive (NAb+, titers ³ 20NU/ml, Group 1) vs. antibody negative (NAb-, titers < 20NU/ml, BAb-, titers <8U, Group 2) patients at the month 6 visit.
2. To compare b-IFN induced biomarker response (viperin, IFIT1) in neutralizing antibody positive (NAb+, titers ³ 20NU/ml, Group 1) vs. antibody negative (NAb-, titers < 20NU/ml, BAb-, titers <8U, Group 2) patients (data compared at baseline and month 6 visits)
3. To compare b-IFN induced biomarker response (MxA, viperin, IFIT1) in neutralizing antibody positive (NAb+, titers ³ 20NU/ml, Group 1) vs. BAb+ (titers ³8U)/NAb- (titers <20 NU/ml, Group 3) patients at baseline and month 6 visits.
4. To correlate NAb titer levels with b-IFN induced biomarker response (data taken from baseline and month 6 visits from Group 1).
5. To compare b-IFN induced biomarker response (MxA, viperin, IFIT1) in BAb-/NAb- patients (Group 2) vs. BAb +/NAb- patients (Group 3) in order to determine if BAbs affect b-IFN induced biomarker response (data compared at baseline and month 6 visits).

Tertiary objectives are:

1. To explore patient characteristics that may predict NAb positivity.

Design: This is a multi-center, open-label study of approximately 300 (200 NAb+ and 100 NAb- (50 BAb+ and 50 BAb-)) MS patients that will compare b-IFN induced biomarker response following b-IFN injection in neutralizing antibody positive vs. antibody negative patients.

Study Population: Approximately 300 subjects (200 in Group 1, 50 in Group 2, and 50 in Group 3) will be recruited for the study.

Inclusion Criteria: To be eligible for entry into this study, candidates must meet all of the following eligibility criteria at the time of randomization:

1. Patients (male or female) diagnosed with relapsing forms of MS.
2. Currently being treated with the same b-IFN (in accordance with FDA approved dosing and schedules) for 12 to 48 months inclusive.
3. All levels of disability
4. Age 18-65 years inclusive
5. Subjects must be willing to be followed for the 6-month study period.

Exclusion Criteria: Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of study initiation.

1. Patients with prior b-IFN NAb test (whether positive or negative).
2. Patients who are currently being treated or have been treated within 6 months prior to screening with combination therapy (b-IFN plus any other immunosuppressant/immunomodulatory) other than IV steroids (either pulse or for a relapse).
3. Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
4. Any other reasons that, in the opinion of the Investigator, the subject is determined to be unsuitable for enrollment into this study.

Treatment Groups: This is a multi-center, open-label study of approximately 300 (200 NAb+ patients and 100 NAb- patients (50 BAb+ and 50 BAb-)) relapsing MS patients that will compare b-IFN induced biomarker response following b-IFN injection in neutralizing antibody positive vs. antibody negative patients.

Subjects currently on any of the three b-IFN preparations (Avonex (Interferon b-1a 30 mcg IM Q 7 days), Rebif (Interferon b-1a 22 or 44mcg SC TIW), or Betaseron (Interferon b-1b 250mcg SC QOD)) will be enrolled to one of 3 groups:

Group 1: Approximately 200 subjects will be enrolled who are NAb+ (titer ³ 20NU/ml)

Group 2: Approximately 50 subjects will be enrolled who are BAb- (titer <8U) and NAb- (titer <20 NU/ml)

Group 3: Approximately 50 subjects will be enrolled who are BAb+ (titer ³8U) and NAb- (titer <20 NU/ml)

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) diagnosed with relapsing forms of MS.
2. Currently being treated with the same b-IFN (in accordance with FDA approved dosing and schedules) for 12 to 48 months inclusive.
3. All levels of disability
4. Age 18-65 years inclusive
5. Subjects must be willing to be followed for the 6-month study period.

Exclusion Criteria:

1. Patients with prior b-IFN NAb test (whether positive or negative).
2. Patients who are currently being treated or have been treated within 6 months prior to screening with combination therapy (b-IFN plus any other immunosuppressant/immunomodulatory) other than IV steroids (either pulse or for a relapse).
3. Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
4. Any other reasons that, in the opinion of the Investigator, the subject is determined to be unsuitable for enrollment into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients on interferon beta
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Eickenhorst, MD, Study Director — Biogen
Locations (28):
- United States (28):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Physicians Resource Network, Cullman, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California - Irvine, Irvine, California
  - University of California San Francisco - MS Center, San Francisco, California
  - Tampa Neurology, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - OSF Saint Francis Medical Center, Illinois Neurological Institute, Peoria, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Mercy Ruan Neurology Clinic, Des Moines, Iowa
  - Kentucky Neuroscience Research / University Neurologists, P.S.C, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - BJC Medical Group, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Family Health Center, White Plains, New York
  - The Multiple Sclerosis Center at the Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University / Rhode Island Hospital, Providence, Rhode Island
  - The Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - The Advanced Neurosciences Institute, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine - The Methodist College Multiple Sclerosis Center, Houston, Texas
  - The University of Texas Houston, Houston, Texas
  - Neurology Center of Fairfax, Ltd., Fairfax, Virginia
  - University of Washington, Seattle, Washington
  - Neurology Associates of Tacoma, Tacoma, Washington